CLINICAL TRIAL: NCT05713019
Title: Neuroinflammatory Interactions of ATP and P2X3 Receptor in the Airways of Chronic Cough Patients: an Exploratory Study
Brief Title: ATP and P2X3 Receptor in Chronic Cough
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Imperial College London (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: IRAS271140
Record Dates: First submitted 2023-01-12; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Cough
Keywords: CHRONIC COUGH; ADENOSINE TRIPHOSPHATE (ATP),; P2X3 receptor
MeSH Terms: conditions — Cough; Chronic Cough

STUDY DESIGN:
Intervention Model Description: Compare effect of diluent with ATP.
Who Masked: Participant, Investigator
Masking Description: Participant and Investigator will be blinded as to whether saline or ATP is being given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effect of saline (Placebo Comparator): Saline will be inhaled from a nebuliser
  Interventions: Device: Adenosine triphosphate (ATP) solution inhalation from nebuliser; Diagnostic Test: Inhalational challenge with increasing concentrations of capsaicin solutions; Device: Recording of Cough Count and frequency using the Hyfe Cough Monitor; Procedure: Collection of exhaled breath condensate; Diagnostic Test: Continuous laryngoscopic examination; Diagnostic Test: Sputum induction; Diagnostic Test: Spirometric measurements; Diagnostic Test: Blood sample collection
- Effect of ATP (Active Comparator): ATP solution will be inhaled from a nebuliser
  Interventions: Device: Adenosine triphosphate (ATP) solution inhalation from nebuliser; Diagnostic Test: Inhalational challenge with increasing concentrations of capsaicin solutions; Device: Recording of Cough Count and frequency using the Hyfe Cough Monitor; Procedure: Collection of exhaled breath condensate; Diagnostic Test: Continuous laryngoscopic examination; Diagnostic Test: Sputum induction; Diagnostic Test: Spirometric measurements; Diagnostic Test: Blood sample collection

INTERVENTIONS:
Device: Adenosine triphosphate (ATP) solution inhalation from nebuliser — ATP and 0.9% saline solution will be inhaled from a nebuliser on separate days, and their effects will be examined.
  Other Names: 0.9% saline solution inhalation from nebuliser
Diagnostic Test: Inhalational challenge with increasing concentrations of capsaicin solutions — Coughs are counted for one minute after single-breath inhalations of 0.9% sodium chloride and capsaicin solutions of increasing concentrations (0.98-500 μm) generated from a dosimeter (P.K. Morgan Ltd, Gillingham, UK) set at a dosing period of 1 s. The concentration that caused more than 2 or 5 coughs was recorded as C2 and C5, and the data is analysed as log10 C2 or C5.
  Other Names: Capsaicin cough challenge
Device: Recording of Cough Count and frequency using the Hyfe Cough Monitor — All enrolled study participants will be provided with a dedicated Android phone or watch loaded with the Hyfe Research application to monitor and record their cough sounds. The participant will be provided with a carrying case to ensure the phone stays within five feet of their mouth. They will be asked to "wear" the phone for the duration of 3 weeks, and keep the phone within five feet of their mouth over nights - keeping it, i.e., on a bedside table.
  Hyfe is a research use only tool which does not provide clinical diagnosis. Cough collection within this study will not lead to specific medical interventions or differential clinical management. Hyfe records only short snippets (<0.5 seconds). As such, the recordings will not be identifiable. Conversations or acoustic environments are not recorded. The informed consent form will explicitly describe exactly what is recorded.
Procedure: Collection of exhaled breath condensate — EBC will be collected by asking the subject to breathe normally onto a handheld breath collection apparatus from Respire Diagnostics, Imperial College, that will cool the exhaled breath to allow for condensation of the exhaled air. The subject will breathe for 2 periods of 5 minutes each separated by a 3-4 min rest to allow the collection of up to 500 uL of liquid. The liquid will be stored for later analysis.
Diagnostic Test: Continuous laryngoscopic examination — Continuous laryngoscopy testing is performed based on previous methodology. Continuous laryngoscopy testing is performed by placing a fibreoptic nasendoscope in the posterior nasopharynx and securing it using specialist headgear. A small quantity of lubricating jelly is used to ease passage of the scope. Video images of the laryngeal inlet are, thereafter, continuously recorded whilst a subject performs various manoeuvres including respiratory movements and cough. These movements will be observed and recorded before and following the various aspects of the challenge protocol and thus allow us to evaluate laryngeal movement abnormalities and for example position of the vocal folds. The size and change in size of the glottic aperture will be evaluated.
Diagnostic Test: Sputum induction — Sputum is induced by inhalation of an aerosol of sterile 3% saline solution and subsequently increasing to 4% and 5% during 3 periods of 5 minutes each. Particular care is taken to avoid contamination with saliva and post-nasal drip by instructing subjects to rinse orally with water and to blow their nose after each inhalation. Sputum samples are collected into sterile pots. Peak flow measurements are made after each inhalation. If there is a fall in peak flow of 20% or more or if symptoms occurred during the procedure, the induction is stopped.
  Sputum plugs are selected and one portion is used to perform differential cell counts. To perform differential cell counts, dithiothreitol is added to the sputum plug and mixed vigorously on a plate shaker to solubilize the sputum. Cytospins are then prepared, and differential cell counts obtained.
Diagnostic Test: Spirometric measurements — Spirometry (FEV1 and forced vital capacity, FVC) is measured using a dry wedge spirometer (Vitalograph, Buckinghamshire, UK).
Diagnostic Test: Blood sample collection — Venous blood (30 cc) will be taken from a vein in the forearm. This test causes a transient discomfort as a needle is used to obtain the blood sample. The blood sample will be used for measuring various proteins and for getting white blood cells to obtain some types of stem cells.

SUMMARY:
This is a laboratory-based study that will be performed at the Clinical Research Centre at the Royal Brompton Hospital,London. The objectives are:

1. Determine whether adenosine triphosphate (ATP) is present or released in airways of idiopathic chronic cough patients
2. Determine whether there is an increase in cough sensitivity and laryngeal sensitivity to exogenous ATP
3. Examine the effects of exogenous ATP on the inflammatory response in the upper and lower airways.

The participants will be: (i) Healthy subjects: non-smoker (8 subjects) and (ii) Chronic cough subjects attending Chronic Cough clinic (12 subjects). Each will be involved in:

Study 1. Following recruitment, subjects will attend for a fiberoptic bronchoscopy.

Study 2: Subjects will take part in a study of the effect of inhaling nebulized ATP. Subjects will be studied on 2 days separated by at least 5 days. On each day, after measurements of lung function, FeNO and cough questionnaires, the subject will inhale either saline or ATP solution from a nebulizer, following which laryngeal hypersensitivity, capsaicin cough challenge and sputum induction will be performed.

Results will be expressed as mean ± standard error of the mean (SEM). Study data will be analysed by the Investigators at the completion of the study. Planned analyses will be done by comparing chronic cough patients to the healthy controls. The Spearman rank-correlation test will be used to determine correlations.

DETAILED DESCRIPTION:
These are the objectives of this study:

1. Determine whether ATP is present or released in airways of idiopathic chronic cough patients
2. Determine whether there is an increase in cough sensitivity and laryngeal sensitivity to exogenous ATP
3. Examine the effects of exogenous ATP on the inflammatory response in the upper and lower airways.

Outcome measures

These are all primary outcome measures of this study:

1. Presence of ATP in airways of idiopathic chronic cough patients and the localisation of P2X2/3 receptors in the airways
2. Cough sensitivity and laryngeal sensitivity to exogenous ATP
3. Inflammatory response in the upper and lower airways to exogenous ATP.

Study Design Consent will be obtained prior to screening. Screening: Participants will be screened prior to engagement in Studies. Normal non-coughing patients will be asked whether they have a history of cough and they should not have had a chronic cough for 8 weeks or more. Those participants with chronic cough need to satisfy the definition of a chronic cough having lasted for more than 8 weeks. These participants will be recruited from the Royal Brompton Hospital Cough clinic. We will use the inclusion and exclusion criteria noted below with regard to eligibility confirmation.

Study 1 and 2 Participants will be in this research project for a total of 3 months.

This study will be in two parts which may not be chronological in order:

Study 1. Following recruitment, subjects will attend for a fiberoptic bronchoscopy.

Study 2: Subjects will take part in a study of the effect of inhaling nebulized ATP. Subjects will be studied on 2 days separated by at least 5 days. On each day, after measurements of lung function, FeNO and cough questionnaires, the subject will inhale either saline or ATP solution from a nebulizer, following which laryngeal hypersensitivity, capsaicin cough challenge and sputum induction will be performed. The order of the ATP or saline challenge will be randomized and the administration of either will be blinded to the patients and investigators measuring the response to the challenge.

Subject population:

This will be a single site study. The investigators will recruit 12 patients with chronic cough attending our Cough Clinic at the Royal Brompton Hospital and 8 control healthy subjects (age and gender matched).

The participants of either gender with idiopathic chronic cough will be studied and should have had a chronic cough of at least 8 weeks' duration, and should have been followed in the Cough Clinic for at least 6 months. These participants will have undergone a protocol with a diagnostic pathway as recommended by the European Respiratory Society guidelines for management of cough. Participants would have either an identifiable cause for their cough that have failed therapies targeted towards the identified cause or classed as having chronic idiopathic cough where no identifiable cause has been found.

The control non-coughing subjects will be recruited through advertisement within the hospital and local newspaper services.

Research Intervention and procedures Fiberoptic bronchoscopy Bronchoscopy is a standard diagnostic procedure and will be undertaken by an experienced doctor of the research team.

The fibre-optic bronchoscope will be passed through either the nasal passages or the oropharynx before passing into the trachea. The nasal passages will be the preferential route, but in case this cannot be done through the nasal passages, the oropharynx will be used. Bronchoalveolar lavage (BAL) will be performed from the right middle lobe using warmed 0.9% saline with 4 successive aliquots of 60ml. The bronchoscopist will then take samples of the cells lining the airways using a brush and forceps, the latter allowing small pieces of tissue to be obtained.

Post-procedure, the participant will be moved from the procedure room to the recovery area, where he/she will be monitored by nursing staff. In case of any bronchoconstriction, he/she will be treated with nebulized salbutamol, and if required, corticosteroid therapy will be given. Once stable, and no longer requiring oxygen and no longer drowsy, he/she will be discharged following review by the research doctors. The doctor may however determine that you need to be kept under observation until fit to be discharged home. Any patient given midazolam during the procedure will be asked to have a responsible adult to accompany them home on that day.

Local anaesthetic is used prior to the procedure and participants may experience a numb mouth or throat. In some patients, if safe to do so, an anxiolytic drug (midazolam) will be given in small doses through the cannula. This is usually tolerated without problem.

After the procedure participants may experience a sore throat, hoarse voice or cough due to irritation to the airways, but this usually settles within a few hours. Other symptoms can include the increased production of sputum, sometimes with blood streaking of the mucus and a transient fever which can occur after a few hours after the procedure. This usually settles within a few hours and can be helped by taking paracetamol. There should be no long-lasting sequelae.

Serious risks are rare but include a pneumothorax (1 in 2000 cases) and significant bleeding. Participants will be closely monitored following the procedure and should any serious complication arise, they will be given the appropriate treatment in hospital.

Exhaled breath condensate (EBC) collection. EBC will be collected by asking the subject to breathe normally onto a handheld breath collection apparatus from Respire Diagnostics, Imperial College, that will cool the exhaled breath to allow for condensation of the exhaled air. The subject will breathe for 2 periods of 5 minutes each separated by a 3-4 min rest to allow the collection of up to 500 microlitre (uL) of liquid. The liquid will be stored for later analysis.

Blood sample collection Venous blood (30 cc) will be taken from a vein in the forearm. This test causes a transient discomfort as a needle is used to obtain the blood sample. The blood sample will be used for measuring various proteins and for getting white blood cells to obtain some types of stem cells.

Continuous laryngoscopic examination Continuous laryngoscopy testing is performed based on previous methodology. Continuous laryngoscopy testing is performed by placing a fibreoptic nasendoscope in the posterior nasopharynx and securing it using specialist headgear. A small quantity of lubricating jelly is used to ease passage of the scope. Video images of the laryngeal inlet are, thereafter, continuously recorded whilst a subject performs various manoeuvres including respiratory movements and cough. These movements will be observed and recorded before and following the various aspects of the challenge protocol and thus allow us to evaluate laryngeal movement abnormalities and for example position of the vocal folds. The size and change in size of the glottic aperture will be evaluated.

Capsaicin cough challenge Capsaicin challenge is performed as established in our laboratory.

The Leicester Cough Questionnaire. This will be used to assess the impact of chronic cough on the patients' quality of life.

Measurement of cough frequency Cough frequency will be measured objectively with a Hyfe cough recording monitor for 48 hours.

All enrolled study participants will be provided with a dedicated Android phone or watch loaded with the Hyfe Research application to monitor and record their cough sounds.

Cough recording will include 5 solicited coughs at the time of study enrolment for calibration. Study personnel will have the ability to remotely monitor the accrual of coughs for each participant in real time with the Hyfe Research Platform Dashboard - thus verifying as needed that the phones are on and functioning appropriately.

Upon study completion, a trained study staff member will retrieve the phones and ensure that data has been automatically uploaded to the Hyfe server.

Assessment of laryngeal function by questionnaire We will use the Laryngeal Hypersensitivity Questionnaire for assessing laryngeal dysfunction.

Induction of sputum Sputum is induced by inhalation of an aerosol of sterile 3% saline solution and subsequently increasing to 4% and 5% during 3 periods of 5 minutes each. Sputum samples are collected into sterile pots.

Sputum plugs are selected and one portion is used to perform differential cell counts. To perform differential cell counts, dithiothreitol is added to the sputum plug and mixed vigorously on a plate shaker to solubilize the sputum. Cytospins are then prepared, and differential cell counts obtained.

In addition, some of the cells will be placed in RNA later for RNAseq analysis. The supernatant will be kept for later assay of neuroimmune biomarkers.

Spirometric measurements Spirometry (FEV1 and forced vital capacity, FVC) is measured using a dry wedge spirometer (Vitalograph, Buckinghamshire, UK).

Fractional exhaled nitric oxide (FeNO) Fractional exhaled nitric oxide (FeNO) level is measured using a portable FeNO monitor (NObreath; Bedfont Scientific Ltd, Rochester, UK) at a constant expiratory flow of 0.05 L/s.

Specimens from bronchoscopy (i) Bronchial brushings: (a) slides with cells attached will be obtained and preserved for later immunohistochemical analysis (b) cells will be placed in RNA later for later extraction for RNAseq analysis (c) cells will be placed in culture.

(ii) Bronchial biopsies: Five μm sections will be cut and stained with haematoxylin and eosin to assess morphology. Investigators will measure the extent of inflammation and remodeling in these biopsies as previously described. In addition, these sections will be used for a series of immunohistochemical investigations for localization of ATP and other associated neuroimmune biomarkers of interest.

(iii) Bronchoalveolar lavage: Bronchoalveolar lavage cells will be placed in cytospin for counting of differential cells. Some of the cells will be kept in RNAlater for RNAseq. The supernatant BAL fluid will be kept for later assay of neuroimmune markers including ATP.

ELIGIBILITY:
Inclusion Criteria:I

1. For Normal non-smoking subject:

   Healthy individuals, free of significant disease No history of asthma/rhinitis, No therapies, Baseline FEV1 ≥80% predicted with FEV1/FVC ratio >70% Non-smoker for at least the past 12 months with a pack history of ≤5 pack-years
2. For chronic cough participants:

   History of chronic cough of at least 8 weeks' duration and should have been followed in the Cough Clinic for at least 6 months.

   Undergone a protocol with a diagnostic pathway as recommended by the ERS guidelines for management of cough.

   Would have either an identifiable cause for their cough that have failed therapies targeted towards the identified cause or classed as having chronic idiopathic cough where no identifiable cause has been found.
3. General Inclusion Criteria:

Give written informed consent prior to participation in the study including all of its procedures.

Comply with the requirements and restrictions listed in the consent form. Male or female subject aged between 30 and 70 years old at screening. Able to complete the study and all measurements. Able to read, comprehend, and write at a sufficient level to complete study related materials.

Exclusion Criteria:

1. General exclusion criteria:

   Subjects will not be eligible if any of the following apply: -
   * As a result of medical interview, physical examination or screening investigation the investigators consider the subject unfit either because of risk to the subject due to the study or the influence this may have on the study results.
   * A history of recreational drug use or allergy which in the opinion of the investigators contra-indicates their participation.
   * Female who is pregnant or lactating or up to 6 weeks post-partum or 6 weeks cessation of breast feeding at any point in the study.
   * Any participants who are involved in current research or have recently been involved in any research prior to recruitment.
   * Those, in the opinion of the investigator, who may prove non-compliant with study procedures.
   * History of an upper or lower respiratory infection (including coryza) within 3 weeks of baseline assessments (assessments and entry could be deferred).
   * Persons who might not adequately understand verbal explanations or written information given in English, or who have special communication needs.
   * Subjects who are currently involved in other research.
2. Specific exclusion criteria for patients with chronic cough:

   1. Exclusion of chronic cough patients with a clear history of asthma and Chronic obstructive pulmonary Disease (COPD) on maintenance therapy
   2. Subjects who are current smokers or ex-smokers with a greater than 10 pack-year history of smoking
   3. Subjects with significant presence of airflow obstruction with an FEV1 of <70% of predicted for age and gender.
   4. Significant vocal cord disorder (VCD).
   5. Long term antibiotic treatment or receipt of a course within 4 weeks of bronchoscopy.
   6. Diagnosis of Allergic bronchopulmonary aspergillosis (ABPA), Churg-Strauss, rheumatoid arthritis, connective tissue disorders; Angiotensin-converting enzyme inhibitor and beta-blockers treatment.
   7. Morbid obesity (BMI>35).
   8. Non-steroid immunosuppressive treatments including methotrexate.

      -

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-28 (Estimated); Primary Completion 2024-03-28 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Does ATP inhalation compared to that of saline inhalation change capsaicin cough sensitivity and laryngeal sensitivity? | 18 months
  Capsaicin cough sensitivity will be measured as the concentration of capsaicin causing 2 or 5 coughs, ie C2 or C5 concentrations in micromolar units. Laryngeal sensitivity will be measured as the change in the area of the glottic aperture between expiration and inspiration maneouvre.
Compare the levels of ATP in bronchoalveolar lavage fluid and in exhaled breath condensate from chronic cough patients to those of non-coughing healthy subjects | 18 months
  This will be done by measurement of ATP concentration in nanomolar units using an off-line luminometer in broncholaveolar lavage fluid and exhaled breath condensate by a paired analysis.

SECONDARY OUTCOMES:
Determine the number of coughs and cough frequency after ATP and saline inhalation in chronic cough and in non-coughing participants. | 18 months
  Cough frequency (coughs per hour) will be measured on the Hyfe Cough Monitors, and the cough frequency per hour over the first 24 hours will be compared between ATP inhalation and saline inhalation in each group (chronic cough and non-coughing participants).
Does ATP inflammation induce granulocytic inflammation after inhalation of ATP? | 18 months.
  The proportion of the granulocytes, neutrophils and eosinophils, will be counted in the induced sputum samples after inhalation of ATP or saline, and the % of neutrophils and eosinophils after ATP or saline inhalation will be compared in each of the 2 participant groups. These measurements will be done from slides on which the sputum cells have been laid out and the results will be expressed as % of the total number of cells on the slide.

CONTACTS AND LOCATIONS:
Overall Officials: Kian Fan Chung, MD, Principal Investigator — Imperial College London